CLINICAL TRIAL: NCT02061553
Title: Use of SMS Messaging to Promote Emotional Health for People With Traumatic Brain Injury: A Randomized Controlled Trial
Brief Title: SMS Messaging to Reduce Depression and Anxiety Following TBI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Albert Einstein Healthcare Network (Other)
Collaborators: National Institute on Disability, Independent Living, and Rehabilitation Research (U.S. Federal Agency)
Responsible Party: Principal Investigator, Amanda Rabinowitz, Institute Scientist, Albert Einstein Healthcare Network
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: TBIMS HN4473; H133A120037 (Other Grant/Funding Number: NIDRR/U.S. Dept. of Education)
Record Dates: First submitted 2014-02-11; First posted 2014-02-13 (Estimated); Last update posted 2023-10-23 (Actual); Status verified 2023-08

CONDITIONS: Traumatic Brain Injury
Keywords: traumatic brain injury; TBI; head injury; brain injury; depression; anxiety
MeSH Terms: conditions — Brain Injuries, Traumatic; Craniocerebral Trauma; Brain Injuries; Depression; Anxiety Disorders | interventions — Information Motivation Behavioral Skills Model; Intention to Treat Analysis

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Motivation (Sham Comparator): 1 in person session focused on importance of motivation followed by 8 wk SMS messages with self-selected motivational statements.
  Interventions: Behavioral: Motivation
- Intention (Active Comparator): 1 session of Behavioral Activation followed by 8 wk SMS messages in the form of BA- based implementation intentions.
  Interventions: Behavioral: Intention
- BA-Tech (Experimental): 6 in person and 2 phone sessions of Behavioral Activation with EMA-based activity monitoring and SMS-assisted scheduling of value-based activities.
  Interventions: Behavioral: BA-Tech

INTERVENTIONS:
Behavioral: Motivation — Control condition in which participants receive a single session with education on the importance of self-confidence and motivation, followed by 8 weeks of daily SMS messages with self-selected motivational statements.
  Arms: Motivation
Behavioral: Intention — Implementation intentions are created collaboratively by participants and therapists in a single 2-hour session that uses principles of brief BA (the planning of rewarding activities). BA-based implementation intentions will then be delivered daily by text for 8 weeks.
  Arms: Intention
Behavioral: BA-Tech — Participants undergo a total of 8 sessions with a therapist. During these sessions, participants learn about the principles of BA (the translation of important life values into the planning of rewarding activities that support those values). The participants' values are explored and an activity schedule is created collaboratively by participants and therapists based on those values. Reminders to complete the scheduled activities will then be delivered by text once the schedule is made. Participants in this arm will also be monitoring their daily activities (and rating them based on enjoyment and perceived achievement) using a cell phone application.
  Arms: BA-Tech

SUMMARY:
This investigation addresses emotional health in community dwelling persons with traumatic brain injury (TBI). It is designed to test the efficacy of a novel behavioral treatment for depression and anxiety symptoms. This treatment incorporates principles of Behavioral Activation (BA), a promising treatment model for depression and anxiety after TBI, and implementation intentions, a theoretically motivated method to enhance enactment of goal-relevant behaviors via action planning. To maximize the impact of this intervention over time, we use the low-cost, widely available technology of SMS, or text messaging, to promote positive behavior change in accordance with planned values and intentions. Participants are randomized 1:2:2 to one of three conditions. Condition 1: a control condition in which participants receive SMS messages with self-selected motivational statements. Condition 2: a condition using BA-based implementation intentions. Condition 3: a condition using BA-based activity monitoring and scheduling based on personal values.

DETAILED DESCRIPTION:
This study employs a 3-group randomized controlled design to examine the efficacy of treatment based on BA using SMS (i.e., text messages) containing reminders to perform scheduled activities based on personal values. These activities are determined collaboratively by participants and therapists during therapy sessions using principles of BA, which incorporates the translation of important life values into the planning of rewarding activities that support those values.

Participants will be randomized 1:2:2 to one of three conditions. The first is a control condition in which participants receive a 2-hour session with education on the importance of self-confidence and motivation, followed by 8 weeks of daily SMS messages with self-selected motivational statements (Motivation group). The second condition uses BA-based implementation intentions delivered daily x 8 weeks (Intention group). The third condition (BA-Tech) has a total of 8 therapy sessions, 6 in person and 2 by phone, and uses BA-based activity scheduling with SMS reminders, plus app-based ecological momentary assessment (EMA) for monitoring the relations among activities, contexts, and reward. The first condition will control for non-specific motivating effects of attention from a therapist and the novelty or "alerting" value of receiving SMS messages. The second condition introduces the idea of Behavioral Activation but does not contain activity monitoring or value-based activity scheduling.

Participants in the Motivation and Intention groups will be contacted by phone at 4 weeks to offer modifications or replacements for their messages. Participants in the BA-Tech group will be able to modify their messages weekly once begun. We will compare groups on change over 8 weeks on: (1) emotional status, (2) perceived degree of environmental reward, (3) degree of behavioral activation, (4) societal participation, and (5) satisfaction with life.

ELIGIBILITY:
Inclusion Criteria:

* TBI (open or closed), sustained at least 6 months prior, of at least complicated-mild injury severity as evidenced by loss or alteration of consciousness not due to intoxication/ sedation and/ or positive neuroimaging findings consistent with TBI;
* At least mild depression and/ or anxiety as evidenced by a score of >5 on PHQ-9 and/ or GAD-7, but without endorsement of suicidal ideation
* Independent in basic home activities and able to travel independently in the community
* Fluent in English and able to communicate adequately for participation in the experimental protocol

Exclusion Criteria:

* History of serious mental illness such as schizophrenia, schizo-affective disorder, or well-documented bipolar disorder;
* Current psychiatric instability, including very severe depression/ anxiety as indicated by PHQ-9 or GAD-7 ≥20; current substance dependence; or active suicidal ideation
* Significant cognitive disability for reasons other than TBI (e.g., developmental disability);
* Inability to use phone texting function due to sensory or motor limitations;
* Concurrent involvement in one-to-one counseling or psychotherapy for emotional issues.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 119 (Actual)
Dates: Start 2013-10-22 (Actual); Primary Completion 2023-05-09 (Actual); Study Completion 2023-07-13 (Actual)

PRIMARY OUTCOMES:
Change from baseline on Brief Symptom Inventory-18 (BSI-18) Global Severity Index | Baseline, 8 weeks (post-treatment)
  The Brief Symptom Inventory (BSI) measure consists of 18 emotional distress items that are rated on a 5 point Likert scale and yield a Global Severity Index as well as Symptom Dimensions (Somatization, Depression, Anxiety.

CONTACTS AND LOCATIONS:
Overall Officials: Amanda Rabinowitz, PhD, Principal Investigator — Moss Rehabilitation Research Institute
Locations (1):
- Moss Rehabilitation Research Institue, Elkins Park, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Hart T, Vaccaro M, Collier G, Chervoneva I, Fann JR. Promoting mental health in traumatic brain injury using single-session Behavioural Activation and SMS messaging: A randomized controlled trial. Neuropsychol Rehabil. 2020 Sep;30(8):1523-1542. doi: 10.1080/09602011.2019.1592761. Epub 2019 Mar 14. PMID 30870102